CLINICAL TRIAL: NCT02990637
Title: The Effect of Olive Leaf Extract Administration on Cardiovascular Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Yala Stevens, MSc., Maastricht University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 163004
Record Dates: First submitted 2016-12-09; First posted 2016-12-13 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Overweight and Obesity; Elevated Cholesterol
Keywords: Olive leaf extract; Cardiovascular health; Cholesterol
MeSH Terms: conditions — Overweight; Obesity; Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- OLECOL (Active Comparator): Olive leaf extract
  Interventions: Dietary Supplement: OLECOL
- Placebo (Placebo Comparator): Maltodextrin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: OLECOL — Olive leaf extract
  Arms: OLECOL
Dietary Supplement: Placebo — Maltodextrin
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effects of daily supplementation of OLECOL for a period of 8 weeks on cardiovascular risk markers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals
* Age between 18 and 70 years
* Total cholesterol levels ≥ 5.0 mmol/L
* BMI 25-35 kg/m2

Exclusion Criteria:

* History of severe cardiovascular, respiratory, urogenital, gastrointestinal/hepatic, hematological/immunologic, HEENT (head, ears, eyes, nose, throat). Dermatological/connective tissue, musculoskeletal, metabolic/nutritional, endocrine, neurological diseases, allergy, major surgery and /or laboratory assessments that might limit participation in or completion of the study protocol.
* Diabetes
* Use of medication that might have influence on endpoints (e.g. cholesterol lowering medication, hypertension medication)
* Administration of investigational drugs or participation in any scientific intervention study which may interfere with this study in the 180 days prior to the study
* Use of antibiotics in the 30 days prior to the start of the study
* Use of antioxidants, minerals and vitamin supplements available in pharmacies, drugstores, food markets or in alternative medicine
* Pregnancy, lactation
* Abuse of products (> 20 alcoholic consumptions per week and drugs)
* Smoking
* Weight gain or loss (> 3 kg in previous 3 months)
* High physical activity (>4.5 hours of running/week)
* History of any side effects towards intake of olives

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-06; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Blood lipid profile | 8 weeks

SECONDARY OUTCOMES:
Lipid peroxidation | 8 weeks
Glucose metabolism | 8 weeks
Systolic and diastolic blood pressure | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ad Masclee, MD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands

REFERENCES:
- [Derived] Stevens Y, Winkens B, Jonkers D, Masclee A. The effect of olive leaf extract on cardiovascular health markers: a randomized placebo-controlled clinical trial. Eur J Nutr. 2021 Jun;60(4):2111-2120. doi: 10.1007/s00394-020-02397-9. Epub 2020 Oct 9. PMID 33034707